CLINICAL TRIAL: NCT03036956
Title: The Prevalence of Sub Clinical Hypothyroidism During Early Pregnancy in Pakistan
Acronym: PRECIOUS
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Dimension Research (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIDI051
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Subclinical Hypothyroidism
Keywords: subclinical hypothyroidism in pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Precious study is likely to help determine the frequency (percentage) of subclinical hypothyroidism among pregnant women in Pakistan It will also help to determine the risk factors for developing subclinical hypothyroidism during pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be enrolled into the study
* Patient between 18-45 years of age; is pregnant and in First Trimester
* Patient willing to give blood sample for laboratory testing
* Patient willing to provide written authorization to obtain data for the study
* Exclusion Criteria:
* Patients suffering from any

  * Chronic Cardiac Disease - Chronic Cardiac Failure, Cardiac Arrhythmia
  * Hepatic Disorder : Cirrhosis
  * Renal Disease : Patients on dialysis and Transplant Therapy
  * Respiratory Disorder
* Subjects with history of non-thyroid malignancy
* Patient currently taking medication for hyperthyroidism
* Active systemic infection
* Patient with physical or mental impairment
* Patients on systemic steroid therapy or lithium therapy
* Patients in second or third trimester of pregnancy
* Patient not willing to give blood sample for laboratory testing
* Patient not willing to provide written authorization to obtain data for the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary Care Clinic/Private Clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Frequency of subclinical hypothyroidism in pregnant females | 12 months
  Continuous variables with normal and non-normal distributions would be reported as mean (SD) and median [inter-quartile range (IQR)], respectively. Prevalence of subclinical hypothyroidism with 95% confidence Interval (CI) will be calculated. Continuous variables between group will compared by using Independent sample t test, and categorical variables will compare by using the chi-square test.

SECONDARY OUTCOMES:
The risk factors that might be associated with subclinical hypothyroidism in all enrolled pregnant patients. | 12 months
  Odds Ratios (OR) and their 95% Confidence Intervals (CI) will be estimated using Logistic Regression. The likelihood ratio test used to assess the association between the explanatory variables and the risk of the subclinical hypothyroidism. Univariable analyses will perform to examine the effect of each variable on the risk of subclinical hypothyroidism. In multivariate analysis all insignificant variables (p >0.05) will check for their confounding and interaction effects before their removal from the final model.

CONTACTS AND LOCATIONS:
Overall Officials: Raeefuddin Ahmed, MD, Study Director — Abbott
Locations (9):
- Pakistan (9):
  - Isra University hospital, Hyderābād
  - Pakistam Insititute of Medical science, Islamabad
  - Atia Hospital Hospital, Karachi
  - Boluvard Hospital, Karachi
  - MediCell Hospital, Karachi
  - Services Hospital, Lahore
  - Sir Ganga Ram hospital, Lahore
  - Welcare Medical Centre, Muzafferabad, Azad Kashmir
  - Lady Reading hospital, Peshawar

IPD SHARING:
Plan to Share IPD: No